CLINICAL TRIAL: NCT06022458
Title: Prenatal Sonographic Prediction of Placental Histology and Function
Status: Recruiting | Type: Observational
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Sunitha Suresh, Physician, FPA, Endeavor Health
Other Study IDs: EH23-068
Record Dates: First submitted 2023-08-08; First posted 2023-09-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy Complications
Keywords: placenta pathology; adverse pregnancy outcomes
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this two-phase observational study is to investigate the use of ultrasonography to predict placental pathology at the time of delivery.

DETAILED DESCRIPTION:
Placenta pathology is examined at the time of delivery and can show the underlying pathophysiology of adverse pregnancy outcomes. The Amsterdam consensus has identified four primary categories of injury, acute inflammation, fetal vascular malperfusion, maternal vascular malperfusion, and chronic inflammation associated with adverse obstetric outcomes. Findings from placental pathologic examination performed at delivery can reveal important patterns of injury that lead to adverse pregnancy outcomes but cannot aid in preventing these outcomes. Ultrasound of the placenta may be able to detect placental pathology in the antepartum period to potentially aid in detection and treatment of placental injury. One specific scenario it may be useful in is in the setting of fetal growth restriction, which can be constitutional or pathologic. Identification of growth restriction in the setting of placental injury may identify those patients at greatest risk for adverse outcomes.

In the retrospective portion of this study, researchers will retrospectively evaluate archived ultrasonographic images during pregnancies affected by stillbirth, severe placental histology, fetal growth restriction, and milder histologic abnormalities. The goal of this phase is to develop image processing of placentas and to utilize the image processing of existing sonograms to correlate with the presence or absence of placental pathology at the time of delivery.

The prospective portion of this study the researchers will utilize image processing techniques from the initial phase to prospectively assess placental function. The goal of this phase is to evaluate if placental size, vasculature, and echogenicities among fetuses with suspected growth restriction are associated with maternal vascular mal perfusion on placental pathology. Twenty patients with fetal growth restriction by estimated fetal weight (EFW) < 10th percentile or fetal abdominal circumference (AC) < 10th percentile and EFW < 20th percentile will be recruited as the exposure group. Participants who consent will complete sonographic measurements of the placenta, predefined image capture of color flow to the placenta, and grayscale images every two weeks. Another twenty patients without SGA (small for gestational age) or significant comorbidities will be recruited in the unexposed control group. Upon consenting, these participants will complete sonographic measurements of the placenta for one time. For both groups, information will be abstracted from electronic medical records regarding demographic data, neonatal outcomes, and placental histology. Imaging characteristics will be compared by placental histology and grade of histology at delivery. As this is a pilot project, there is not an a priori power analysis.

ELIGIBILITY:
Retrospective Phase

Inclusion criteria:

* Patients with delivery in NorthShore University HealthSystem,
* Ultrasound available within 4 weeks of delivery with adequate placental images
* Placental pathology available

Exclusion criteria:

* Multiple gestation

Prospective Phase Inclusion criteria

* Exposed: Patients with singleton gestation with fetal growth restriction at 20-28 weeks with a plan to deliver at NorthShore Highland Park Hospital Evanston Hospital. Patients must have a first-trimester ultrasound (<14 weeks) to confirm pregnancy dating available in the electronic medical record.
* Unexposed: Patients who present for routine ultrasound evaluation at 36-38 weeks with normal fetal growth with a plan to deliver at NorthShore Highland Park Hospital or NorthShore Evanston Hospital.

Exclusion criteria:

* Exposed: Multiple gestation, major fetal anomaly
* Unexposed: Multiple gestation, history of chronic hypertension, gestational or pregestational diabetes, major fetal anomaly antiphospholipid syndrome, known thrombophilia

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only patients of the female sex will be recruited and a large majority will identify as female.
Study Population: Pregnant patients who plan to deliver at NorthShore University HealthSystem
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Imaging characteristics | Image characteristics will be collected every 2 weeks prenatally, and placenta will be collected at the time of delivery for analysis, this will be up to 22 weeks
  Imaging characteristics will be compared by those with and without placental pathology found at the time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Sunitha Suresh, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided